CLINICAL TRIAL: NCT02146417
Title: A Phase IV, Blinded, Randomized Controlled Trial to Compare the Effectiveness of Low Pressure Pneumoperitoneum - With Profound Muscle Relaxation - During Laparoscopic Donor Nephrectomy to Optimize the Quality-of-recovery During the Early Post-operative Phase
Brief Title: Comparison of Low Versus Normal Pressure Pneumoperitoneum - With Profound Low Versus Normal Pressure Pneumoperitoneum -With Profound Muscle Relaxation- During Laparoscopic Donor Nephrectomy
Acronym: LEOPARD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISP#51414
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Renal Disease
Keywords: Low pressure pneumoperitoneum; Deep neuromuscular block
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal pressure pneumoperitoneum & deep neuromuscular block (Active Comparator): Normal pressure pneumoperitoneum
  Interventions: Procedure: Normal pressure pneumoperitoneum (12 mmHg); Procedure: Deep neuromuscular block
- Low pressure pneumoperitoneum & deep neuromuscular block (Experimental): Low pressure pneumoperitoneum
  Interventions: Procedure: Low pressure pneumoperitoneum; Procedure: Deep neuromuscular block

INTERVENTIONS:
Procedure: Low pressure pneumoperitoneum
  Arms: Low pressure pneumoperitoneum & deep neuromuscular block
Procedure: Normal pressure pneumoperitoneum (12 mmHg)
  Arms: Normal pressure pneumoperitoneum & deep neuromuscular block
Procedure: Deep neuromuscular block

SUMMARY:
As both patients with end-stage kidney disease and society benefit tremendously from live kidney donation, the safety and well-being of kidney donors are highly important objectives in live kidney donation. Laparoscopic donor nephrectomy has several advantages over open nephrectomy, such as less post-operative pain, better quality of life and shorter hospital stay. Therefore, laparoscopic donor nephrectomy is nowadays the treatment of choice in most countries.

So far, modifications of the technique of laparoscopic donor nephrectomy, i.e. hand-assisted and/or retroperitoneoscopic approaches, did not show a significant benefit with regard to safety as reflected by the conversion to open and postoperative complications rate. We therefore believe that further research should focus on the optimization of early postoperative pain and its concomitant use of opioids. Since non-steroidal anti-inflammatory drugs are contra-indicated before and after nephrectomy, the management of postoperative pain largely depends on the administration of opioids. Measures to reduce postoperative pain would also reduce the occurrence of postoperative nausea and vomitus, and postoperative bowel dysfunction.

A recent pilot study performed by our group showed that the use of low pressure pneumoperitoneum was feasible and significantly reduced deep intra-abdominal and referred pain score during the first 72 hours after surgery. Previous studies performed by others show that low pressure pneumoperitoneum is associated with reduction of systemic inflammatory response, post-operative pain and analgesic consumption. Martini et al have shown that deep neuromuscular block improves surgical conditions during laparoscopic surgery with standard intra-abdominal pressure. To facilitate the use of low pressure pneumoperitoneum, deep neuromuscular block improves surgical conditions and might become a prerequisite for the use of low pressure pneumoperitoneum.

Our hypothesis is that the combination of low pressure pneumoperitoneum and deep neuromuscular block improves quality of recovery in the early post-operative phase.

ELIGIBILITY:
Inclusion Criteria:

* obtained informed consent
* age over 18 years

Exclusion Criteria:

* insufficient control of the Dutch language to read the patient information and to fill out the questionnaires
* chronic use of analgesics or psychotropic drugs
* use of non-steroidal anti-inflammatory drugs shorter than 5 days before surgery
* known or suspect allergy to rocuronium or sugammadex
* significant liver* or renal** dysfunction
* neuromuscular disease
* pregnant of breastfeeding
* indication for rapid sequence induction

  * liver dysfunction is defined as alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) > twice the upper limit (extremely rare in live kidney donors) ** renal dysfunction is defined as serum creatinine twice the normal level and/or glomerular filtration rate < 60 ml/min (extremely rare in live kidney donors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality-of-Recovery 40 scale | day 1

SECONDARY OUTCOMES:
Cumulative use of opioids | Day -1;0;1;2;3 and Mon3
Cumulative use of other analgetics | Day -1;0;1;2;3
Post-operative complications | Day 0;1;2;3 and Month 3
Time to reach discharge criteria | Day 0;1;2;3

OTHER OUTCOMES:
Operation time | Peri-operative
Length of pneumoperitoneum | Peri-operative
Estimated blood loss | Peri-operative
Intra-operative complications | Peri-operative

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Warlé, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Reijnders-Boerboom GTJA, van Helden EV, Minnee RC, Albers KI, Bruintjes MHD, Dahan A, Martini CH, d'Ancona FCH, Scheffer GJ, Keijzer C, Warle MC. Deep neuromuscular block reduces the incidence of intra-operative complications during laparoscopic donor nephrectomy: a pooled analysis of randomized controlled trials. Perioper Med (Lond). 2021 Dec 9;10(1):56. doi: 10.1186/s13741-021-00224-1. PMID 34879862
- [Derived] Albers KI, van Helden EV, Dahan A, Martini CH, Bruintjes MHD, Scheffer GJ, Steegers MAH, Keijzer C, Warle MC. Early postoperative pain after laparoscopic donor nephrectomy predicts 30-day postoperative infectious complications: a pooled analysis of randomized controlled trials. Pain. 2020 Jul;161(7):1565-1570. doi: 10.1097/j.pain.0000000000001842. PMID 32107359
- [Derived] Ozdemir-van Brunschot DMD, Scheffer GJ, van der Jagt M, Langenhuijsen H, Dahan A, Mulder JEEA, Willems S, Hilbrands LB, Donders R, van Laarhoven CJHM, d'Ancona FA, Warle MC. Quality of Recovery After Low-Pressure Laparoscopic Donor Nephrectomy Facilitated by Deep Neuromuscular Blockade: A Randomized Controlled Study. World J Surg. 2017 Nov;41(11):2950-2958. doi: 10.1007/s00268-017-4080-x. PMID 28608013
- [Derived] Ozdemir-van Brunschot DM, Scheffer GJ, Dahan A, Mulder JE, Willems SA, Hilbrands LB, d'Ancona FC, Donders RA, van Laarhoven KJ, Warle MC. Comparison of the effectiveness of low pressure pneumoperitoneum with profound muscle relaxation during laparoscopic donor nephrectomy to optimize the quality of recovery during the early post-operative phase: study protocol for a randomized controlled clinical trial. Trials. 2015 Aug 12;16:345. doi: 10.1186/s13063-015-0887-7. PMID 26265279